CLINICAL TRIAL: NCT02778607
Title: PROgressive Supranuclear Palsy CorTico-Basal Syndrome Multiple System Atrophy Longitudinal Study UK
Acronym: PROSPECT-M
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University of Cambridge (Other); University of Oxford (Other); University of Manchester (Other); Newcastle University (Other); University of Sussex (Other); Royal Gwent Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14/0371
Record Dates: First submitted 2016-04-22; First posted 2016-05-20 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Progressive Supranuclear Palsy (PSP); Corticobasal Degeneration; Multiple System Atrophy (MSA)
Keywords: Atypical Parkinsonism Syndrome (APS)
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Blood sample collection for: DNA extraction, Peripheral blood lymphocyte storage, plasma, serum and RNA storage.
  2. Brain MRI scan
  3. Skin biopsy
  4. Cerebro-spinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Progressive Supranuclear Palsy: Patients with a current clinical diagnosis of Progressive Supranuclear Palsy (PSP)
- Multiple System Atrophy: Patients with current clinical diagnosis of Multiple System Atrophy (MSA).
- Atypical Parkinsonian Syndrome: Atypical Parkinsonian Syndrome (APS) patients who do not fulfil existing criteria for PSP/CBD/MSA, but may represent variant clinical syndromes related to tau pathology including pure akinesia with gait freezing (PAGF), PSP-parkinsonism, overlap syndromes and atypical parkinsonian disorders not meeting clinical diagnostic criteria at entry
- Controls: Participants unaffected by neurological or psychiatric disease
- Corticobasal Degeneration: Patients with a current clinical diagnosis of Corticobasal Degeneration (CBD)

SUMMARY:
Progressive Supranuclear Palsy (PSP), Cortico-Basal Degeneration (CBD) and Multiple System Atrophy (MSA) are degenerative brain conditions for which there are currently no curative treatments. To aid the development of new treatment trials, there is a pressing need to develop better methods for diagnosing these conditions early, and to track disease progression. The PROSPECT-M-UK study will collect standardised clinical data over time. Patients will also have the option to have a brain MRI scan, eye movement exam and donate blood, skin and spinal fluid samples, with the aim to identify "biomarkers" that can improve the accuracy of early diagnosis and track the natural time course of disease. Control participants and those not meeting criteria for Parkinson's disease or other defined conditions but are considered by the investigator group to be allied syndromes or at risk states (atypical parkinsonian syndromes), will also be examined. Patients can also participate via the CBD European registry or in a one-off study assessment through the cross-sectional study, which involves completing questionnaires and a blood sample donation.

DETAILED DESCRIPTION:
There are a group of neurodegenerative disorders which are often initially diagnosed to be Parkinson's disease (PD), but which are biologically and clinically distinct, and follow a malignant disease course. The three most common conditions are PSP, CBD and MSA. These conditions have a median survival of approximately 6-7 years and unlike PD, do not respond well to dopamine replacement therapy.

PSP and CBD are characterized by tau-pathology and MSA by alpha-synuclein pathology. A great deal of pre-clinical work has been carried out on tau and alpha-synuclein disease models, yet there are no disease modifying agents for these conditions. There are a number of potential therapeutic compounds in development and in order to improve the likelihood of their success, there is a pressing need to increase the number of early case patients recruited into these new treatment trails. Thus, better methods for improved accuracy of early diagnosis and for tracking progression need to be developed. This can be achieved through:

1. a detailed study of the change in patients' clinical state over time;
2. studying "biomarkers" such as blood, skin, spinal fluid and brain MRI.

The investigators will recruit patients with PSP, CBD and MSA who are referred to specialist clinics for assessment and treatment. An additional group of Atypical parkinsonian syndrome (APS) cases who do not meet criteria for Parkinson's disease or other defined conditions, but are considered by the investigator group to be allied syndromes or at risk states will also be invited to participate in the study. People unaffected by neurological disease will be invited to participate on a one-off occasion.

Being involved in the PROSPECT-M-UK longitudinal study will involve attending a research assessment on 5 occasions over 3 years in our natural history cohort, and for 2 occasions over 2 years for our longitudinal cohort. Study procedures consist of: having a neurological examination; completing questionnaires to provide details of clinical history, self/carer reported functional scales and quality of life; neuropsychology assessment; eye movement exam; donating blood and skin samples; some patients will be invited to have a lumbar puncture for spinal fluid collection and have a brain MRI scan on two occasions (at baseline and after 1 year follow-up). Patients can also agree to be contacted by phone or at a clinic appointment for remote monitoring of symptoms after face to face visits have completed.

In addition, a cross-sectional cohort will be established, to enable participation of patients who cannot travel to a study centre. This will involve donating blood samples,returning study questionnaires, and being monitored remotely. A CBD European registry will also be created which will involve a structured neurological assessment, a medical notes review and blood sample donation.

The primary outcome for the study is duration of disease, with the aim to improve methods for early diagnosis and tracking disease progression. Importantly, the study will link together centres and researchers from across Europe to establish the infrastructure and create a trial ready cohort for future therapeutic study into PSP/CBD/MSA.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent obtained prior to any study-related procedures. A consultee process will be used where participants lack the mental capacity for consent, either due to cognitive or communication deficits.
* 2. Fulfills clinical criteria (PSP, MSA, CBD/CBS) or clinically defined allied disorders (at-risk states or intermediate disorders, as above) or a healthy control participant recruited from local volunteer databases or next of kin where they have expressed a wish to participate.
* 3. Participant is 18 years old or older.
* 4. Participant has an identified informant.

Exclusion Criteria:

* 1. Participant has another significant medical or psychiatric illness that would interfere in completing assessments
* 2. Participant is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient recruitment for the natural history and longitudinal study arms will be through identification of patients by their physicians. The patients will have been referred or will be receiving treatment at a movement disorders, neurology or medical clinic. Patient recruitment for the cross-sectional study will be i.) through identification of patients attending relevant specialist neurology clinics ii.) through information placed on patient organization websites, PSP Association and MSA Trust, and iii.) patients with CBD/CBS can also be recruited via the British Neurological Surveillance Unit (BNSU).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2014-10; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Survival status after 5 years of clinical follow-up | 5 years
  To determine patient survival status after 5 years of follow-up for survival analysis using the Kaplan-Meier Method

SECONDARY OUTCOMES:
Annual change in degree of disability in PSP, CBD and APS cases as determined by the PSP rating scale | 3 years
  Change in clinical symptoms and motor function in PSP, CBD and APS cases to determine degree of disability and rate of disease progression using a 0-100 rating scale
Annual change in degree of disability in MSA cases as determined by the Unified Multiple System Atrophy Rating Scale (UMSARS) | 3 years
  Change in clinical symptoms and motor function in MSA cases to determine degree of disability and rate of disease progression with scores ranging from 0 to 104

OTHER OUTCOMES:
CSF biomarkers | 1 year
  Changes in CSF biomarkers of neurodegeneration after one year of follow-up including: neurofilament light chain, total tau, tau isoforms, phosphorylated tau
Brain MRI | 1 year
  Whole and regional brain atrophy (%/year) and functional connectivity measured across distinct brain regions (using low frequency BOLD signal) will be examined after 1 year of follow-up using brain MRI.
MoCA Cognitive function test | 3 years
  Cognitive function will be reviewed annually for 3 years using the Montreal Cognitive Assessment (MoCA). The total score is out of 30 with higher scores indicating better cognitive functioning.
ACE-3 Cognitive function test | 3 years
  Cognitive function will be reviewed annually for 3 years using the Addenbrookes Cognitive Examination (ACE-3). The total score is out of 100 with higher scores indicating better cognitive functioning.
ECAS Cognitive function test | 3 years
  Cognitive function will also viewed annually for 3 years using the Edinburgh Cognitive and Behavioural ALS Screen (ECAS). The total score is out of 136 with higher scores indicating better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Huw Morris, PhD, FRCP, Principal Investigator — University College, London
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following the first 2 years of the study a data and samples access committee will be established comprised of a representative of each study site together with representatives of the PSP Association and MSA trust, and will be chaired by an independent member who is experienced in the review of sample and tissue requests. The availability of tissue and samples will be publicized by the PSP Association and MSA trust.